CLINICAL TRIAL: NCT03736473
Title: A Phase I, Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of MEDI9447 (Oleclumab) in Japanese Patients With Advanced Solid Malignancies
Brief Title: A Phase I Study of MEDI9447 (Oleclumab) in Japanese Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D6070C00006
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-06

CONDITIONS: Advanced Solid Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEDI9447 monotherapy (Other): Dose escalation of MEDI9447 monotherapy for patients with advanced solid malignancies
  Interventions: Drug: MEDI9447 (oleclumab)

INTERVENTIONS:
Drug: MEDI9447 (oleclumab) — MEDI9447 administered intravenously

SUMMARY:
This is a phase I, open-label study to assess the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of MEDI9447 in Japanese patients with advanced solid malignancies.This study consists of 2 cohorts. Cohort 1 (dose level 1) and Cohort 2 (dose level 2). At least 3 or up to 6 evaluable Japanese patients with advanced solid malignancies will be enrolled in each cohort.

DETAILED DESCRIPTION:
Objectives:

Primary objective:

To assess the safety and tolerability, describe any dose-limiting toxicity (DLT) for MEDI9447

Secondary objective:

To determine the pharmacokinetics (PK) characteristics of MEDI9447 To determine the immunogenicity of MEDI9447 To evaluate candidate biomarker of MEDI9447 activity in archival tumor biopsy specimens To describe the preliminary antitumor activity of MEDI9447

Exploratory Objective:

To explore profile of biomarker status, with MEDI9447 treatment

Overall design:

This is a phase I, open-label study to assess the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of MEDI9447 in Japanese patients with advanced solid malignancies.

This study consists of 2 cohorts. Cohort (dose level 1) and Cohort 2 (dose level 2).

At least 3 or up to 6 evaluable Japanese patients with advanced solid malignancies will be enrolled in each cohort. The total number of subjects will depend upon the available data in each cohort and Safety Review Committee (SRC)'s decision.

Study Period:

The study is expected to start in October 2018 and end in July 2019.

Number of Subjects:

Maximum 12 evaluable patients will be enrolled in this study.

Treatments and treatment duration:

Subjects will receive MEDI9447 on Day 1 and Day 15 in a 4-week cycle. Subjects participating in the study may continue to receive study treatment(s) as long as they are continuing to show clinical benefit, as judged by the Investigator, unless the subject has progressive disease (PD) with either clinical deterioration and/or no further benefit from treatment, experiences unacceptable toxicity, or should discontinue for any other reason. In such cases, the Investigator needs to consult with the sponsor and they agree to continue study treatment in advance.

Statistical methods:

The primary objective of this study is to assess the safety and tolerability profile of MEDI9447.

All safety data will be summarized using the safety analysis set (All subjects who received at least 1 dose of MEDI9447). Evaluations of safety and tolerability will include, but not be limited to, AEs, physical examinations, laboratory findings (including clinical chemistry, hematology, and urinalysis), vital signs (including blood pressure and pulse), and electrocardiograms using summary statistics.

For secondary and exploratory efficacy endpoints, all analyses will be descriptive, and no formal statistical testing will be performed. Data will be summarized and plotted appropriately according to data type.

PK concentration data for MEDI9447 will be listed for each subject and each dosing day, and summary statistics will be tabulated. Immunogenicity results will be listed by subject, and summaries of the number and percentage of subjects who develop detectable antidrug antibodies (ADAs) against MEDI9447 will be provided. The immunogenicity titre will be listed for samples confirmed positive for the presence of ADAs. Neutralizing ADAs may be reported for samples confirmed positive for the presence of ADAs.

All analyses and reporting will be conducted for each cohort.

ELIGIBILITY:
Major Inclusion Criteria:

* Adult subjects; age ≥ 20 years
* Has a histologically confirmed solid malignancy that is refractory to standard therapy or for which no standard of care regimen currently exists
* Subjects must have at least 1 lesion that is measureable using RECIST v1.1
* All subjects must consent to provide archived tumor specimens for biomarker studies
* ECOG Performance Status of 0 or 1
* Life expectancy ≥12 weeks
* Adequate organ function
* Body weight ≥ 35 kg

Major Exclusion Criteria:

* Patients must have completed any previous cancer-related treatments before enrollment.
* Prior treatment with CD73 antagonist, tumor necrosis factor receptor superfamily agonists
* All CTLA-4, PD-1, or PD-L1 antagonists related-AEs must have resolved to ≤ NCI CTCAE v4.03 Grade 1 or baseline prior to screening and not worsened before the first dose of study drug
* Must not have required the use of additional immunosuppression other than corticosteroids for the management of an CTLA-4, PD-1, or PD-L1 related AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day
* Known allergy or hypersensitivity to the study drug, its compounds, or agents similar biologic composition
* History of more than one event of IRR requiring permanent discontinuation of IV drug treatment
* History of severe drug allergies or anaphylaxis to 2 or more food products or medicine
* Cardiac or peripheral vascular disease
* NCI CTCAE v4.03 Grade 3 or greater edema
* Uncontrolled massive ascites or pleural effusion
* History of NCI CTCAE v4.03 Grade 3 or greater thromboembolic events within 3 months prior to the first dose of study drug or thromboembolic event of any grade with ongoing symptoms
* Active tuberculosis
* Patients with history of, or current ILD
* Active or prior documented autoimmune within the past 3 years prior to the start of treatment
* Untreated or unstable CNS metastatic disease, leptomeningeal disease, or cord compression
* Concurrent enrollment in another clinical study
* Any concurrent chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment
* Toxicities from prior anticancer therapy that have not resolved to ≤ NCI CTCAE v4.03 Grade 1 or baseline prior to the first dose of study drug
* History of primary immunodeficiency or solid organ transplantation
* Active hepatitis B, hepatitis C, or HIV
* Females who are pregnant, lactating, or intend to become pregnant during their participation in the study
* Other invasive malignancy within 2 years prior to the first dose of study drug
* Uncontrolled concomitant illnes
* Judgment by the Investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions, and requirements.
* Involvement in the planning and/or conduct of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Adverse event | From the informed consent to 90 days after the last dose
  To assess the safety and tolerability, describe any dose-limiting toxicity (DLT) for MEDI9447

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Chūōku, Japan